CLINICAL TRIAL: NCT03990467
Title: Observed Pharmacokinetic of Piperacillin/Tazobactam in ICU Patients Compared to Therapeutic Drug Monitoring of Amikacin
Brief Title: Observed Pharmacokinetic of Piperacillin/Tazobactam Compared to Amikacin in ICU
Acronym: OPTIMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0843
Record Dates: First submitted 2019-06-04; First posted 2019-06-19 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Septic Shock; Sepsis; Sepsis Syndrome
MeSH Terms: conditions — Shock, Septic; Sepsis; Systemic Inflammatory Response Syndrome | interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated by amikacin and piperacillin (Experimental): ICU patient with a sepsis treated by amikacin and piperacillin/tazobactam
  Interventions: Biological: Plasma dosage of amikacin, piperacillin and tazobactam

INTERVENTIONS:
Biological: Plasma dosage of amikacin, piperacillin and tazobactam — Pharmacokinetic (PK) criteria will be used to judge whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam

SUMMARY:
The pharmacokinetics of antimicrobials is profoundly modified in Intensive care unit (ICU) patients. To adapt the treatment, it is recommended to measure blood levels of antibiotics. Some antibiotics, such as amikacin, are easy to monitor, while for other molecules, such as piperacillin/tazobactam, the drug monitoring is more difficult to obtain. These two molecules have similar physicochemical characteristics (hydrophilicity) and therefore have closed pharmacokinetic properties. OPTIMA is a study aiming at criteria will be used to judge whether the pharmacokinetic (PK) parameters of amikacin are predictive of those of piperacillin and tazobactam.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient hospitalized in the critical care department of the Lyon-Sud hospital centre
* Patient with a sepsis or a severe sepsis table defined by the latest international recommendations
* Patient to be treated by the amikacin + piperacillin/tazobactam association
* Patient affiliated to a social security system, having agreed to participate in the study

Exclusion Criteria:

* Patient with a known history of hypersensitivity or contraindication to amikacin, piperacillin or tazobactam
* Patient known to have previously received piperacillin/tazobactam or amikacin combination before inclusion
* Patient treated at the time of inclusion with dialysis techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-01-28 (Estimated); Study Completion 2023-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in plasma concentration of amikacin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
Change in plasma concentration of piperacillin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
Change in plasma concentration of tazobactam during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
Dose administered of amikacin at baseline | Hour 0 (Baseline)
Dose administered of piperacillin at baseline | Hour 0 (Baseline)
Dose administered of tazobactam at baseline | Hour 0 (Baseline)
Change in plasma volume of distribution of amikacin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma volume of distribution is one of the two PK parameters evaluated in this study (with clearance), calculated with drug plasma concentration and dose administered
Change in plasma volume of distribution of piperacillin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma volume of distribution is one of the two PK parameters evaluated in this study (with clearance), calculated with drug plasma concentration and dose administered
Change in plasma volume of distribution of tazobactam during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma volume of distribution is one of the two PK parameters evaluated in this study (with clearance), calculated with drug plasma concentration and dose administered
Change in plasma clearance of amikacin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma clearance is one of the two PK parameters evaluated in this study (with volume of distribution), calculated with drug plasma concentration and dose administered
Change in plasma clearance of piperacillin during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma clearance is one of the two PK parameters evaluated in this study (with volume of distribution), calculated with drug plasma concentration and dose administered
Change in plasma clearance of tazobactam during the first 24 hours after administration | First 24 hours of the antimicrobial treatment (Hour 1, Hour 5, Hour 7 and Hour 24)
  In order to evaluate whether the PK parameters of amikacin are predictive of those of piperacillin and tazobactam.
  Plasma clearance is one of the two PK parameters evaluated in this study (with volume of distribution), calculated with drug plasma concentration and dose administered

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie et Réanimation - Secteur de Soins Critiques, Groupement Hospitalier Sud, HCL, Pierre-Bénite, France